CLINICAL TRIAL: NCT06210802
Title: Validation of Korean Version of Defense and Veterans Pain Rating Scale (DVPRS) for Assessment of Postoperative Pain
Brief Title: Validation of K-DVPRS
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2311-172-1489
Record Dates: First submitted 2023-12-28; First posted 2024-01-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Korean version of Defense and Veterans Pain Rating Scale — Defense and Veterans Pain Rating Scale translated into Korean

SUMMARY:
This study aimed to validate Korean version of Defense and Veterans Pain Rating Scale for the assessment of postoperative pain.

DETAILED DESCRIPTION:
Defense and Veterans Pain Rating Scale (DVPRS) is translated into the Korean version through forward-back translation. The K-DVPRS is reviewed by the Korean expert and finally verified by the investigator of this study.

On a day before surgery, postoperative pain at rest and during cough is investigated using K-DVPRS, and K-DVPRS supplementary questions and EQ-5D-5L are conducted. At 24 hours after surgery, postoperative pain of surgical site at rest and during cough is investigated using NRS and K-DVPRS, and K-DVPRS supplementary questions and EQ-5D-5L are conducted. At this time, to assess the reliability of K-DVPRS, postoperative pain of surgical site at rest and during cough is re-investigated using K-DVPRS after 30-60 minutes. At 48 hours after surgery, postoperative pain of surgical site at rest and during cough is investigated using NRS and K-DVPRS, and K-DVPRS supplementary questions and EQ-5D-5L are conducted.

In order to verify the reliability of the K-DVPRS, the internal correlation coefficient (ICC) and Cronbach's alpha coefficient are calculated to evaluate the test-retest reliability. Convergent validity and construction validity are calculated to verify the validity of the K-DVPRS. Spearman correlation analysis between pain intensity at rest and during cough using NRS and K-DVPRS is performed to verify convergent validity. In addition, an inter-item correlation analysis is conducted between pain intensity at rest and during cough using K-DVPRS, scores of K-DVPRS supplemental questions, pain intensity at rest and during cough using NRS, and EQ-5D-5L scores. To verify the construct validity, K-DVPRS score is analyzed by age, sex, operation time, and the severity of surgery. Finally, the Mann-Whitney U test is used to compare the difference in postoperative during at rest and during cough evaluated by K-DVPRS before and 24 hours after surgery. The difference in postoperative pain between 24 and 48 hours after surgery is also compared in the same way. The evaluation success rates of NRS and K-DVPRS are also compared at postoperative 24 and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic surgery or robot abdomen surgery (duration ≥ 1 hour) under general anesthesia

Exclusion Criteria:

* Patients with ASA PS ≥ III
* Patients with a difficulty to answer postoperative pain-related questions or K-DVPRS
* Patients with red-green color blindness or difficulty distinguishing colors
* Patients who are inappropriate for this clinical trial based on the investigator's opinionr

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic surgery or robot abdomen surgery (duration ≥ 1 hour) under general anesthesia in Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Validity of K-DVPRS | at postoperative 24 and 48 hours
  convergent validity and construct validity
Reliability of K-DVPRS | at postoperative 24 hours
  test-retest reliability

SECONDARY OUTCOMES:
Evaluation success rate of K-DVPRS | at postoperative 24 and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No